CLINICAL TRIAL: NCT02809807
Title: The Impact of the Work of Breathing and Gas Exchange for COPD Patient Using a Gas Mask.
Brief Title: Gas Mask and Chronic Obstructive Pulmonary Disease (COPD): New Understanding on the Respiratory Index Impact?
Acronym: COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Captain (retired) Stephane Bourassa, RN CD (Unknown); Mr Pierre-Alexandre Boucard, RT (Unknown)
Responsible Party: Principal Investigator, François Lellouche, Research Director, Laval University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: 21140MPOC
Record Dates: First submitted 2016-06-20; First posted 2016-06-22 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Work of Breathing
Keywords: Work of Breathing; Hypoxemia; Respiratory Acidosis; Respiratory effort; COPD
MeSH Terms: conditions — Hypoxia; Acidosis, Respiratory; Pulmonary Disease, Chronic Obstructive | interventions — Respiratory Protective Devices

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Baseline (Experimental): Without a gas mask. We measure baseline respiratory index, parameters and the comfort.
  Interventions: Other: measurement of the work of breathing
- Assessment with gas mask and canister A (Experimental): With a gas mask, the measurement have been done with a high resistive canister. We measure baseline respiratory index, parameters and the comfort. These would serve for conduction comparison with the baseline.
  Interventions: Other: measurement of the work of breathing; Device: Gas Mask
- Assessment with gas mask and canister B (Experimental): With a gas mask, the measurement have been done with a low resistive canister. We measure baseline respiratory index, parameters and the comfort. These would serve for conduction comparison with the baseline.
  Interventions: Other: measurement of the work of breathing; Device: Gas Mask

INTERVENTIONS:
Other: measurement of the work of breathing — We have been evaluating breathing patterns, index of respiratory efforts and blood gases in all randomized conditions. Airway pressure, inspiratory and expiratory flows have been measured. An esophageal catheter has been introduced at the beginning of the study to measure esophageal pressure (Peso) and calculate indexes of respiratory effort (PTPeso, WOB). SpO2 has been continuously measured and capillary blood bases were drawn at the end of each condition. Comfort has also been assessed. FreeO2 System has been used and pre-programmed in accordance with the patient SpO2 target zone for potential correction of the hypoxemia occurrences. Differences among randomized conditions are one without gas mask as for the baseline and two with gas masks but different canisters.
Device: Gas Mask — Differences among randomized conditions are one without gas mask as for the baseline and two with gas masks but different canisters.
  Other Names: Canadian Gas Mask (C4, Airboss Defence, Bromont, Canada) and Canisters (C7A1 and ABD81)
  Arms: Assessment with gas mask and canister A; Assessment with gas mask and canister B

SUMMARY:
Background: The gas mask is used to protect the aiways against respiratory hazards (CBRN agents). Within the CBRNE committee, speculations are that unprotected lungs would look like to those of COPD patients in post-exposure of some CBRNE agents. The aim of the study was to evaluate the impact of the gas mask on respiratory patterns and indexes of the respiratory effort. Methods: We are completing our study with 9 COPD patients to evaluate breathing patterns, index of respiratory efforts and blood gases. Three conditions have been tested in a randomized order: 1x baseline and 2x different canisters, with and without a mask (C4, Airboss Defence, Bromont, Canada). Airway pressure, inspiratory and expiratory flows have been measured. An esophageal catheter is introduced at the beginning of the study to measure esophageal pressure (Peso) and calculate indexes of respiratory effort (PTPeso, WOB). SpO2 is continuously measured and capillary blood bases are drawn at the end of each condition. Each condition lasts 10 minutes, data of the last 2 minutes at a steady state are considered for analyses. Results. We are compiling data and processing them for analysis.

DETAILED DESCRIPTION:
The principal way of penetration of CBRNE agents is the respiratory system. The current technology of a gas mask has been used to protect the respiratory system as far back as the First World War. That originated from Dr Cluny Macpherson's initiatives whom was a Canadian military physician.

The military gas mask is part of the respirator classification but owes its specific features. Conventionally, the military gas mask covers a large spectrum of protection aspects and matched with their specific canisters. Consequently, gas masks are usually studied separately from other respirators and Self-Contained Breathing Apparatus (SBCA). While few studies have been about the gas mask technology, no-study addresses it in regards of the impact from a bad airway protection and consequences on the respiratory system.

The gas mask design and its components may lead to these respiratory load issues. At rest and from different resistances, what would be the impacts for the work of breathing and gas exchange? In order to avoid hypoxemia and hyperoxia, what would be the optimal means to restore proper oxygenation? We hypothesised on a: i. Heightened WOB and the respiratory demands related to wear of the gas mask; ii. An occurrence of hypoxemia will be manifesting during a continuous period. Our goal is to measure the impact of the work of breathing and the gas exchange for a gas mask user and also a COPD patient. We also measure what was the optimal means for correcting the hypoxemia with a subject.

9 COPD patients have been participating in a comparison and single-blind randomized experimental study. That was approved by the Ethical Review Committee. A written consent is obtained for all the subjects prior their acceptance. No rejection has happened during the recruiting so far. The eligibility criteria are: i. COPD diagnosis from mild-to-severe FEV 30-80%). The exclusion criteria are: i. Refusals relate to wear the oesophageal catheter and for capillary punctures; ii. Claustrophobia; iii. Oesophageal wounds backgrounds; iv. No coronary background and stroke history; v. No face morphology incompatibility with the mask. Spirometry and usual health screening is also done before starting the clinical trial.

Design comprises three 10-minute testing conditions split in two parts. All has been at rest and sitting on a chair: i. Baseline without gas mask; ii. Gas mask and Canister A; iii. Gas Mask and Canister B. Between the condition a 5-minute wash-out takes place.

Three five-minute periods is followed to record blood pressure and pulse during the conditions. SpO2 is continuously measured with Free O2. Capillary punctures are done at the end of each condition. Comfort was also assessed.

Our main measurements are the WOB performed with a continuous recording of Peso pressure and respiratory volumes. Software Acknowledge, version 3.9 serves as acquisition data system and analysis are achieved with a 4.2 version and a free-trial WOB calculus system, named RESPMAT. That is obtained from Maynaud and al.(2014). As power source, we use a BIOPAC (MP100, Santa Barbara, Californie, USA, 200 Hertz), four differential sensors (Validyne : 1x MP45±100 cmH2O; 2x MP100±5 cmH2O; 1x MP100±100 cmH2O) and four Carrier D-Modulators (Validyne, CT-15,120 Volt, 60 Hertz, 5Watts, Model CD15-A-2-A-1).

Single esophageal catheter (Type Cooper, French caliber #5) and disposable pneumotachs are used. Lidocain spray and K-Y gel are applied during the insertion of the catheter. Its placement is done at 37.6±5.7 cm across the subject and a Mueller test is performed for each subject. In regard of spontaneous breathing, an Hudson mask is used while a C-4 Gas Mask with a canister was employed (Manufacturer: Airboss Defence, Bromont, Canada). Canister A and B were respectively a C7A1 and ADB81 trademark. Prototyped Free O2 System is employed for the correction of the hypoxemia.

ELIGIBILITY:
Inclusion Criteria:

• COPD Diagnosis: mild-to-moderate, with FEV1 30-80% and requiring no long-term oxygenotherapy.

Exclusion Criteria:

* Refuse to participate in the study for one of the following reasons: i. wearing a oesophageal catheter; ii. wearing the gas mask; iii. giving blood sample; iv. claustrophobia.
* Oesophageal background wounds
* Facial anthropometrical issues.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Indexes of respiratory effort | 10 minutes
  At rest

CONTACTS AND LOCATIONS:
Overall Officials: Francois Lellouche, PhD, Principal Investigator — Laval University
Locations (1):
- Institut de Recherche Universitaire de Cardiologie et Pneumologie de Québec, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bourassa S, Bouchard PA, Dauphin M, Lellouche F. Oxygen Conservation Methods With Automated Titration. Respir Care. 2020 Oct;65(10):1433-1442. doi: 10.4187/respcare.07240. Epub 2020 Feb 18. PMID 32071135